CLINICAL TRIAL: NCT03957447
Title: Treat Early and Broad: Thermotherapy of Buruli Ulcer Integrated Into WHO-recommended Wound Management in West Africa
Acronym: WOUNDCARE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Centre Suisse de Recherches Scientifiques en Cote d'Ivoire (Other); Institut Pasteur de Côte d'Ivoire, Abidjan Cocody CHU, Côte d'Ivoire (Unknown)
Responsible Party: Principal Investigator, Martin Koch, Medical Writer/Data Entry Supervisor, University Hospital Heidelberg
Other Study IDs: WOUNDCAREV2
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Skin Ulcer; Buruli Ulcer; Nontuberculous Mycobacteria
Keywords: skin wounds; Ivory Coast community health services; prevalence study; thermotherapy
MeSH Terms: conditions — Skin Ulcer; Buruli Ulcer; Hyperthermia | interventions — Hyperthermia, Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients exhibiting skin wounds: Within the framework of Taabo HDSS Cross-sectional community and health services surveys are performed before wound management intervention (main study and substudy 1) is implemented (baseline) and are continued at 6 monthly intervals thereafter. Surveys are done door-to-door. All patients with skin lesions (broken skin barrier) are enrolled, lesions are documented with help of a questionnaire and photographic documentation.
- patients identified in the survey and willing to participate: Each patient with a wound will be enrolled. Presumptive clinical diagnosis and empirical treatment, as well wound assessment, will be recorded at enrollment and at each follow-up visit. Additional laboratory testing done within the framework of the local health system will also be recorded.
- patients exhibiting Buruli ulcers < 2cm: Buruli ulcer patients fulfilling inclusion criteria will be offered thermotherapy instead of standard antibiotic treatment. Heat treatment is applied for 42 days plus a safety margin of up to 14 days, if ulcer margins have not fully collapsed and/or induration has not fully subsided. Treatment terminates earlier, if a lesion is completely closed. Thermotherapy will be applied with heat packs twice daily.
  Interventions: Other: thermotherapy (application of heat): This part of the trial is on hold due to the Covid19-pandemia

INTERVENTIONS:
Other: thermotherapy (application of heat): This part of the trial is on hold due to the Covid19-pandemia — Heat treatment is applied for 42 days plus a safety margin of up to 14 days, if ulcer margins have not fully collapsed and/or induration has not fully subsided. Treatment terminates earlier, if a lesion is completely closed. Thermotherapy will be applied with heat packs twice daily.
  Groups: patients exhibiting Buruli ulcers < 2cm

SUMMARY:
The project rolls out combined innovative low-tech thermotherapy with heat packs and WHO recommended wound management in a Buruli ulcer (BU)-endemic district of West Africa. It addresses three key areas of considerable clinical and public health importance in the region:

* to better help people managing the disabling disease BU that primarily affects children in West Africa
* to implement WHO recommended general wound management for all types of wounds with tools available at the peripheral level of the health care system
* to prevent systemic life threatening sequelae (e.g. sepsis and rheumatic fever) and permanent local damage (e.g. motor and sensory disability) by early recognition and treatment of wounds at the community level. The project translates available research findings already validated on the secondary health care level into clinical practice at the periphery (primary health care level). The string of the investigator's previous work from the development of the BU thermotherapy-wound management-package to the proof of its efficacy provides all necessary skills, tools and documents to immediately proceed into practical community application.

Operational endpoints are

* coverage and quality of WHO recommended wound management training of health care personnel at the primary health care level (health posts);
* coverage, success rate and quality of care for patients with BU and other wounds; denominator controlled at health post level and high-quality Health and Demographic Surveillance Systems (HDSS) data.

The project is embedded into a stable multidisciplinary working environment at Côte d'Ivoire, including an HDSS with a longstanding record of partnership and successful community-based operational research.

The project builds on the principles laid out by the Sustainable Development Goals (SDGs) and Universal Health Coverage (UHC) and

* targets all patients with a broken down skin barrier independent of the cause (patient centred health care)
* brings diagnosis and treatment close to the community
* educates and trains both community members and health care workers
* measures the health intervention outcome The project is fully in line with the new integrated strategy for the skin NTDs of WHO's Department of Control of NTDs (WHO/NTD).

DETAILED DESCRIPTION:
Overall goal of the study To contribute to a better understanding of the clinical epidemiology of wounds and wound healing and to improve wound management in settings with limited resources at the community level, the primary and secondary level of the health care services.

Study objectives Main study

* To measure the proportion of wounds healed (defined as wound closed) at each cycle of clinical diagnosis and the corresponding presumptive treatment
* To describe the clinical epidemiology of wounds presented (presumptive clinical and confirmed diagnoses)
* Coverage and quality of wound management training of health care personnel at the peripheral health care level (health posts); Substudy 1
* To measure the effectiveness and acceptability of thermotherapy of patients with early BU (< 2cm) treated at health post level with the following outcomes:

  * Primary endpoints absence of clinically BU specific features' according to WHO guidelines or 'wound closure' within 6 months after completion of heat treatment ("primary cure") and 'absence of BU recurrence for 12 months after completion of heat treatment' ("definite cure").
  * Secondary outcomes rates of withdrawal for low compliance consent withdrawal rating of thermotherapy by health staff Substudy 2
* To measure the frequency and the severity of skin lesions (broken skin barrier) in the community and the health services
* To investigate the determining factors of community and health services-based wound management
* To measure the impact of the wound management intervention (main study and substudy 1) on the frequency, spectrum and severity of wounds including systemic complications in the community and at the 7 health posts / district hospital (HDSS-based) compared to the baseline study before the intervention and over time after the implementation of the intervention.

Target Population The target population are approximately 43,000 people of the Taabo HDSS which is surveyed longitudinally for key demographic, health and socioeconomic indicators since 2008. This provides ideal conditions to implement the intervention and assess the impact through operational endpoints. The health centres and the district hospital involved are part of the public health system. There is one district hospital and the seven health posts within the Taabo DHSS.

ELIGIBILITY:
Inclusion Criteria:

Survey All HDSS population members Wound management study Patients with wounds defined as broken skin barrier. Thermotherapy study Buruli ulcer patients of the main study with ulcers < 2cm.

Exclusion Criteria:

none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in Taabo Health District (HDSS), Ivory Coast Survey All HDSS population members Wound management study Patients with wounds defined as broken skin barrier. Thermotherapy study Buruli ulcer patients of the main study with ulcers < 2cm.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-05-07 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of skin ulcers in inhabitants of the Taabo health district, Ivory Coast | 2 years
  To measure the frequency and the severity of skin lesions (broken skin barrier) in the community and the health services
Qualitative description of factors determining public health services-based skin ulcer managment | 2 years
  Description of facilitating and obstructive factors for recognition and treatment of ulcers (questionnaires, interviews, patient and institution-related documentation of costs)
Frequency and severity of skin ulcers after community health service intervention | 2 years
  To measure the impact of the wound management intervention (main study and substudy 1) on the frequency, spectrum and severity of wounds including systemic complications in the community and at the health posts / district hospital compared To the baseline study before intervention and over time after implementation of the intervention.
Number of patients with healed skin ulcers identified in the survey (see outcome 1) | 2 years
  To measure the proportion of ulcers healed at each cycle of clinical diagnosis and corresponding presumptive treatment
Number of patients presenting at the health posts level with skin ulcers identified in the survey (see above) | 2 years
  To describe the clinical epidemiology of different types of skin ulcers (wounds) presented (presumptive clinical and confirmed diagnoses)
Quality of care for patients with skin ulcers identified in the survey (see above) | 2 years
  Coverage and quality of skin ulcer (wound) management training of health care personnel at the peripheral health care level (health posts)
Outcome of patients with Buruli ulcers < 2cm and willing to participate in thermotherapy study | 2 years
  Number of patients completing thermotherapy exhibiting no more signs of clinically Buruli ulcer (BU) specific features' according to WHO guidelines or 'wound closure' within 6 months after completion of heat treatment ("primary cure") and 'absence of BU recurrence for 12 months after completion of heat treatment' ("definite cure").

SECONDARY OUTCOMES:
Drop out rate of patients with Buruli ulcers < 2cm and willing to participate in thermotherapy substudy | 2 years
  Number of participants of the thermotherapy substudy not included in analysis of healing rate (see outcome 7) due to lack of cooperation or failure to return for assessment
Withdrawal of patients with Buruli ulcers < 2cm and willing to participate in thermotherapy substudy | 2 years
  Number of participants with consent withdrawal
Patients with Buruli ulcers < 2cm and willing to participate in thermotherapy substudy | 2 years
  Rating of skin ulcer thermotherapy by health staff of the Taabo health distric, Ivory Coast, measured by a score based on a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Marija Stojkovic, MD, Principal Investigator — University Hospital Heidelberg, Germany
Locations (1):
- CSRS, Abidjan, Côte d’Ivoire

IPD SHARING:
Plan to Share IPD: Undecided
A RedCap datashare platform is in place already. Individual patient data will be provided anonymised.

REFERENCES:
- [Derived] Toppino S, Koffi DY, Kone BV, N'Krumah RTAS, Coulibaly ID, Tobian F, Pluschke G, Stojkovic M, Bonfoh B, Junghanss T. Community-based wound management in a rural setting of Cote d'Ivoire. PLoS Negl Trop Dis. 2022 Oct 13;16(10):e0010730. doi: 10.1371/journal.pntd.0010730. eCollection 2022 Oct. PMID 36227844
- [Derived] Toppino S, N'Krumah RTAS, Kone BV, Koffi DY, Coulibaly ID, Tobian F, Pluschke G, Stojkovic M, Bonfoh B, Junghanss T. Skin wounds in a rural setting of Cote d'Ivoire: Population-based assessment of the burden and clinical epidemiology. PLoS Negl Trop Dis. 2022 Oct 13;16(10):e0010608. doi: 10.1371/journal.pntd.0010608. eCollection 2022 Oct. PMID 36227839